CLINICAL TRIAL: NCT05132257
Title: Genetic Polymorphism and Retinopathy of Prematurity: Correlation of Clinical Presentations and Severity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202001715A3
Record Dates: First submitted 2021-11-02; First posted 2021-11-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Retinopathy of Prematurity; Genetic Polymorphism
Keywords: Retinopathy of prematurity, genetic polymorphism
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Our approach for SNP selection from candidate genes includes maximum utilization of data available from databases (dbSNP, HapMap) and from our own screening for informative genetic markers. In general, SNP variants for genotyping will be selected from available databases, such as dbSNP. In cases where a candidate gene has not been screened comprehensively and/or where data on allele frequencies is not readily available (estimated in 20-25 out of 50 genes, such as ANG-1, ALK-1, etc.), SNPs will be detected by direct sequencing of 20-40 study subjects. This will allow us to identify all alleles with population frequency >5%, including intronic SNPs, variants from the regulatory regions (mainly promoters), and cSNPs included in open reading frames. Data obtained by direct screening also validates the information extracted from databases, which still contain incomplete information in up to 25% of cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PM No-ROP: Premature without retinopathy of prematurity. Prematurity was defined as birth at < 37 weeks gestation.
- Mild ROP: Prematurity with mild retinopathy of prematurity. ROP not needing treatment. Prematurity was defined as birth at < 37 weeks gestation.
- Severe ROP: Prematurity with type 1 retinopathy of prematurity. Prematurity was defined as birth at < 37 weeks gestation.
  Interventions: Procedure: Severe ROP
- Fullterm: Heathal fullterm.

INTERVENTIONS:
Procedure: Severe ROP — The treatment for ROP was either primary intravitreal injection (IVI) of anti-vascular endothelial growth factor (anti-VEGF) or laser photocoagulation or vitrectomy, and the indication for treatment was type 1 ROP, as defined by the ETROP Study.
  Other Names: Type 1 ROP
  Groups: Severe ROP

SUMMARY:
Study Aim and Goals

1. Evaluate the correlation between genetic polymorphism and ROP development
2. To study the possibility if there are any specific genetic polymorphisms that lead to poor outcome or recurrence of ROP after treatment.

DETAILED DESCRIPTION:
Background:

The preterm neonate, especially the low birth weight infant, is at a greater risk to develop disorders in multiple organ systems because of immaturity. Retinopathy of prematurity (ROP) is a disorder of the developing retina of low birth weight preterm infants that has the potential to lead to blindness. Although the pathogenesis and etiology of ROP remains unclear, many causative factors have been proposed. Vascular endothelial growth factor (VEGF) is an important regulator of angiogenesis in fetal life. In humans, polymorphisms in the VEGF gene have been reportedly associated with proliferative diabetic retinopathy and age-related degeneration. These retinal diseases might share the disease process of vasculopathy with ROP. Besides risk factors specifically associated with preterm birth, the activation of pro-inflammatory cytokines has been suggested to contribute to ROP development. Tumor necrosis factor (TNF)-α is one of the major cytokines in inflammation. Its expression was up-regulated in retinal neovascularization in animal models and proliferative eye diseases in humans. Many researchers suggest that TNF-α may affect retinal angiogenesis and predispose preterm infants for later development of ROP. Recent studies showed the possible correlation between ROP and polymorphism in VEGF (-460 T/C, +936 C/T, -634 G/C, and -2578 C/A), or TNF-α (-308 G/A). However, these studies focused on western populations. In our study, we will analyze the relationships among severity, treatment outcomes, and genetic polymorphism findings in ROP.

Study Aim and Goals

1. Evaluate the correlation between genetic polymorphism and ROP development
2. To study the possibility if there are any specific genetic polymorphisms that lead to poor outcome or recurrence of ROP after treatment.

Study Design Participants: We plan to recruit the children born at Linkou and Taipei branches of Chung Gung Memorial Hospital in 2009-2018, who are willing to undergo series of ophthalmologic examinations.

Study period: April, 2021 to March, 2024. A prospective cohort study Inclusion criteria: All children who were born at Linkou and Taipei branches of Chung Gung Memorial Hospital during the period of 2009 to 2018.

Exclusion criteria: If the parents were not willing to participate the study, or the medical records were not complete, or the follow period was less than 6 months.

Estimated patients' numbers: about 500 babies/3 years Methods: Participants will receive series of ocular exams, including: cycloplegic refractions, strabismus exams, exams of intraocular pressure, slit lamp exam, fundus exam, axial length measurement, etc. After the parent's and the participant's agreement, we will have a blood test of 3 ml and undergo DNA collection (Oragene-DNA; DNA-Genotek, Ottawa, Canada) by study personnel. We will analyze around 10 SNPs from each of candidate genes in our study.

According to patients' previous records and images, subjects will be classified as cases and controls. "Cases" will be infants with severe treatment-requiring ROP (defined as type-1 ROP [zone I, any stage, with plus disease; zone I, stage 3, without plus disease; or zone II, stage 2 or 3, with plus disease] or worse). "Controls" will be full-term babies without other retinal disorder, infants with no ROP or with mild ROP less severe than type-1 ROP, who are within the same birth weight group (e.g., <1000 grams or ≥1000 grams). After matching genetic results and structural outcomes, we will analyze whether any specific genetic polymorphism had higher presentations in treatment-requiring ROP patients. Also, secondary analysis will focus on the difference between recurrent/poor outcome cases and other cases.

Statistical Analysis: Continuous variables will be analyzed with independent-t or paired-t test. One-way ANOVA will be used to compare three or more groups. Ordinal variables will be analyzed with Wilcoxon rank sum test (two independent samples) or Wilcoxon signed rank test (tow paired samples). Categorical variables will be analyzed with Chi-square test or Fisher's exact test. A multivariable logistic regression model will be constructed to assess the association between myopia prevalence and all studied risk factors. P value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born at Linkou and Taipei branches of Chang Gung Memorial Hospital during the study period.

Exclusion Criteria:

1. Parents unwilling to participate in the study
2. Incomplete medical records.
3. Folllow-up period less than 6 months
4. Other ocular diagnosis including glaucoma, cataract, FEVR, etc.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We recruit the children born at Linkou and Taipei branches of Chung Gung Memorial Hospital in the study period, who are willing to undergo series of ophthalmologic examination
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
SNP Selection, Detection, and Genotyping | 2021-2024
  We will analyze around 10 SNPs from each of 53 candidate genes in our study population. Genotyping of 500 selected SNPs will be performed by TaqMan genotyping assays (Applied Biosystems, Foster City, CA) on the 7900HT Fast Real-Time PCR System (384-well platform). Primary outcome comprises frequency of mutations in percentage ratio and risk profile analysis (odds ratio).

CONTACTS AND LOCATIONS:
Overall Officials: Wu WeiChi, M.D., PhD., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Ophthalmology, Chang Gung Memorial Hospital., Linkou District, Taoyuan, Taiwan